CLINICAL TRIAL: NCT06806514
Title: The Relationship Between Upper Extremity Exercise Capacity, Respiratory and Peripheral Muscle Strength and Level of Disability in Individuals With Chronic Low Back Pain
Brief Title: The Relationship Between Upper Extremity Exercise Capacity, Respiratory and Peripheral Muscle Strength in Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2025-02/12
Record Dates: First submitted 2025-02-03; First posted 2025-02-04 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Indıviduals with chronic low back pain

SUMMARY:
The aim of the study was to evaluate the upper extremity exercise capacity of individuals with chronic low back pain and to investigate its relationship with respiratory muscle strength, peripheral muscle strength, chest expansion, pain, disability level, fear of movement and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Being aged 18-65
* Chronic low back pain for at least the last 3 months
* Pain intensity according to Visual Analogue Scale (VAS) ≥3

Exclusion Criteria:

* History of cancer
* Presence of spinal infection
* Presence of rheumatological disorders
* Presence of spinal fracture
* Red flag signs
* Having a psychological disorder
* Presence of spinal surgery
* Having radiculopathy
* Presence of anatomical and congenital abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic low back pain who are being followed up at the Department of Physical Medicine and Rehabilitation at Kirsehir Ahi Evran University will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | 1st day
  It will be assessed by 6 minute pegboard and ring test.
Respiratory muscle strength | 1st day
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using a portable mouth pressure device.
Peripheral muscle strength | 1st day
  Knee extensor, shoulder abductor and hand grip strength will be evaluated with a dynamometer.
Chest expansion | 1st day
  Neutral, deep inspiration and deep expiration circumferences will be measured from the axillary, epigastric and subcostal regions using a tape measure.
Disability level | 1st day
  It will be assessed with Oswestry Disability Index. High scores on the scale indicate the presence and severity of symptoms.

SECONDARY OUTCOMES:
Kinesiophobia | 1st day
  It will be evaluated with the Tampa Kinesiophobia scale.The total score ranges from 17-68, with a score above 37 indicating a high degree of kinesiophobia.
Quality of life | 1st day
  It will be evaluated with the Short Form-12 Quality of Life scale.The subscales rate health from 0 to 100, with 0 indicating poor health and 100 indicating good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)